CLINICAL TRIAL: NCT02712450
Title: Tools Development for Geriatric Emergency Regulation at the Emergency Service Centre, in the Rhône Area
Brief Title: Tools Development for Geriatric Emergency Regulation
Acronym: REGESA
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL14_0449
Record Dates: First submitted 2016-02-16; First posted 2016-03-18 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Emergency Geriatric Care
Keywords: geriatric; emergency; clinical pathway; regulation; SAMU; training
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control group: * Patients included from January 2016 to August 2016
  * Before regulating doctors training course
- Experimental group: * Patients included from January 2017 to August 2017
  * After regulating doctors training course

SUMMARY:
According to surveys, 13% to 20% of the Service Médical d'Urgence (SAMU) centre 15 (French 911) calls concern elderly patients above 75 years of age. For these patients, the clinical pathway should be decided on the basis of the symptomatology described during the call, but also with the gathering of specific data such as medical social and psychological evaluation. These items allow the regulating doctor to assess comorbidity, on-going treatment, psycho-cognitive status, previous hospitalisations, social situation, and patient expectations and needs.

However, data collected in order to assess the situation on the phone and take the orientation decision are mainly limited to the severity of clinical symptoms. Medical, psychological and social aspects are rarely gathered, for several reasons :

* Phone call shortness : emergency calls should be treated quickly
* Regulating doctors are not trained to take in account the specificities or geriatric patients in their decision making. Besides, they are not informed about alternatives to the hospital emergency department, such as "geriatric channel" system.

An observational study was performed in 2012 on 692 calls about elderly patients referred to the SAMU centre 15 during 7 days : 63% of these patients were transferred to an emergency department. Regardless of severe cases "hospital regulation", 55% of the least serious cases ("liberal regulation") were transferred to an emergency department.

Regulation is inadequate to elderly patients for whom 1) the situation assessment and the appropriate decision making require specific items that are not known by regulating doctors, 2) the medical care and the clinical pathway could be improved by the knowledge of on-field "geriatric channel", 3) the emergency department care is particularly long, 4) and could be pernicious to younger patients.

1920 patients will be recruited between January 2016 and August 2017, including a 6 months wash-out in order to train regulating doctors. This training will include geriatric patient's specificities, and geriatric channels. A 12% difference between the 2 groups (before and after the training) is expected, considering a 80% statistical power. The design is a time series experiment.

ELIGIBILITY:
Inclusion Criteria:

* Patient above 75 years olds
* Patient calling for a liberal regulation
* Patient calling between 8 a.m. and 6 p.m. from monday to friday

Exclusion Criteria:

* Patient calling for vital emergency (hospital regulation)
* Patient calling for inter-hospital transport

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients calling SAMU
Sampling Method: Probability Sample
Enrollment: 2279 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients sent to an emergency department | 24 hours after patient's call
  The training course efficiency (which contains specific regulation tools and emergency regulation doctors formation) will be assessed by evaluating the proportion of 75 years old patients and older sent to an emergency department after a liberal regulation.

SECONDARY OUTCOMES:
Duration of the hospital stay in emergency department | 7 days after patient's call
  The training course efficiency on hospital stay duration will be assessed by evaluating the duration of the hospital stay in emergency department, after regulating doctor decision.
Occurence of non-programmed hospitalization in emergency department | 7 days after patient's call
  The training course efficiency on non-programmed hospitalization in emergency department will be assessed by evaluating the occurence of these type of hospitalization one week after call regulation
Geriatric channel utilisation rate | 24 hours after patient's call
  Training course efficiency on the geriatric channel utilization by regulating doctors will be assessed using multiple parameters : geriatric hotline use, intra-hospital geriatric mobile team mobilisation, extra-hospital geriatric mobile team mobilisation, direct hospitalization in geriatric department
Training course feasibility | 24 hours after patient's call
  Training course feasibility will be assessed using multiple parameters : regulation call duration, regulating doctor orientation respect, contact between regulating doctor and physician (GP, geriatric doctor, emergency doctor, geriatric channel)
Medical cost for patient | 7 days after patient's call
Non medical cost for patient | 7 days after patient's call
Training course cost | 7 days after patient's call

CONTACTS AND LOCATIONS:
Locations (1):
- Service Gériatrie - Hôpital Edouard Herriot, Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Foucaud A, Gilbert T, Vincent A, Jomard N, Comte B, Porthault S, Comte G, Theurey O, Gueugniaud PY, Bourelly L, Rabilloud M, Boutitie F, Douplat M, Tassa O, Haesebaert J, Termoz A, Schott AM. Evaluation of a training program for emergency medical service physician dispatchers to reduce emergency departments visits. J Am Geriatr Soc. 2023 Feb;71(2):484-495. doi: 10.1111/jgs.18101. Epub 2022 Nov 1. PMID 36317929